CLINICAL TRIAL: NCT03190083
Title: Efficacy of Digital Breast Tomosynthesis (DBT) in Addition to Standard 2- Dimensional Mammography in Evaluating Extent of Disease in Newly Diagnosed Breast Cancer Patients
Brief Title: Efficacy of Digital Breast Tomosynthesis + Standard 2- Dimensional Mammography in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE6117
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2020-04-10 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: mastectomy; lumpectomy; 3-Dimensional Mammogram; digital breast tomosynthesis
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: The radiologist reviewing the tomosynthesis images will be separate and blinded from the radiologist who reviewed the initial 2-D mammogram
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 3-dimensional tomosynthesis mammogram (Experimental): The patients assigned a Breast imaging-reporting and data system (BIRADS) 5 category at the time of diagnosis and all new diagnosed breast cancer patients, will undergo a separate 2-D plus DBT in addition to the standard 2-D mammogram
  Interventions: Device: 2-dimensional mammogram; Device: digital breast tomosynthesis (DBT)

INTERVENTIONS:
Device: 2-dimensional mammogram — This is standard of care for breast cancer diagnosis. The new breast cancer patients will be scheduled for the mammogram after diagnosis at the time of surgical appointment. The radiologist reviewing the tomosynthesis images will be separate and blinded from the radiologist who reviewed the initial 2-D mammogram.
Device: digital breast tomosynthesis (DBT) — The radiation dose from this/these procedure(s) will be no more than 0.4mSv for a bi-lateral breast tomosynthesis. The new breast cancer patients will be scheduled for the mammogram after diagnosis at the time of surgical appointment. The radiologist reviewing the tomosynthesis images will be separate and blinded from the radiologist who reviewed the initial 2-D mammogram.
  Other Names: 3-dimensional mammogram

SUMMARY:
The purpose of this study is to determine if a 3-dimensional mammogram (DBT) may provide additional information to evaluate the extent of disease and additional findings that would aid in staging a new breast cancer patient. This would impact surgical planning and improve patient outcomes.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of the study is to measure the frequency with which DBT alters the surgical plan to mastectomy versus lumpectomy. Only positive findings, like an additional site of cancer or DCIS, will be taken into account when estimating the frequency of changes to surgical management.

Secondary objectives:

1. To measure the frequency and nature of additional findings like atypical pathology (Atypical ductal/ lobular hyperplasia, papilloma, Lobular carcinoma in situ (LCIS) , requiring surgical intervention).
2. To identify variables on 2D (e.g. dense breasts, architectural distortions, non calcified masses) that might predict which patients would benefit from DBT.
3. To measure the proportion of patients undergoing additional work-up following the DBT, and the subset of these patients with benign findings (i.e. False Positives).

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of breast cancer
* New diagnosis if a previous breast cancer patient with negative surgical margins
* Patients willing to sign a written informed consent form

Exclusion Criteria:

* High risk benign lesions as the primary pathology diagnosis

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with a diagnosis of breast cancer and identifying as female
Enrollment: 16 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Sharma, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-dimensional Tomosynthesis Mammogram
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who went on study
Arm/Group | 3-dimensional Tomosynthesis Mammogram
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  years: 20-29 | 1
  years: 30-39 | 2
  years: 40-49 | 4
  years: 50-59 | 6
  years: 60-69 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which DBT Altered Surgical Plan
Description: Only positive findings, like an additional site of cancer or atypical pathology like Atypical ductal/ lobular hyperplasia, papilloma, DCIS/LCIS (findings requiring surgical intervention), will be taken into account when estimating the frequency of changes to surgical management
Time Frame: At completion of 3-Dimensional mammogram (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | 3-dimensional Tomosynthesis Mammogram
Number analyzed (Participants) | 16
Participants | 0

2. Other Pre Specified Outcome: Variables on 2-Dimensional Mammogram That Might Predict Which Patients Would Benefit From DBT
Time Frame: At completion of 3-Dimensional mammogram (1 day)
Reporting Status: Not Posted

3. Other Pre Specified Outcome: The Proportion of Patients Undergoing Additional Work-up Following the DBT
Time Frame: At completion of 3-Dimensional mammogram (1 day)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Patients Undergoing Additional Work-up Following the DBT With Benign Findings
Time Frame: At completion of 3-Dimensional mammogram (1 day)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During tomosynthesis procedure, up to 1 hour
Arm/Group | 3-dimensional Tomosynthesis Mammogram
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03190083/Prot_SAP_001.pdf